CLINICAL TRIAL: NCT06714513
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Explore the Immunogenicity of the Tuberculosis (TB) Vaccine Candidate QTP101 (ID93+GLA-SE) in Older Adults (Aged 55~74 Years)
Brief Title: ID93+GLA-SE Vaccine Against Tuberculosis in Older Adults Aged 55-74
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Quratis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT-QTP101-007; RS-2024-00337483 (Other Grant/Funding Number: Korea Health Industry Development Institute); 31538 (Other: Ministry of Food and Drug Safety (Republic of Korea))
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- BCG-vaccinated, HIV-negative, QFT-negative and middle-aged adults (55-64) with a low dose of QTP101 (Experimental): This study arm evaluates the safety and immunogenicity of a low dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-negative adults aged 55-64. Participants receive 2 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56. The target population includes individuals without prior TB infection as indicated by the QFT-negative status.
  The primary objective is to assess safety, focusing on adverse events (AEs), and to explore immunogenicity through antibody titers and cytokine responses. Findings will provide critical insights into the vaccine's effects in middle-aged, previously uninfected individuals.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-negative and middle-aged adults (55-64) with a high dose of QTP101 (Experimental): This study arm evaluates the safety and immunogenicity of a high dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-negative adults aged 55-64. Participants receive 10 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56. This group focuses on individuals without prior TB infection, as indicated by their QFT-negative status.
  The primary objective is to assess the safety profile, including adverse events (AEs), and to evaluate the immune response, such as antibody titers and cytokine production. The findings will help determine the vaccine's suitability for middle-aged individuals and guide future dose optimization.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-negative and middle-aged adults (55-64) with the placebo (Placebo Comparator): This study arm serves as a placebo comparator for BCG-vaccinated, HIV-negative, QFT-negative adults aged 55-64. Participants receive intramuscular injections of sterile normal saline (placebo) on Day 0, Day 28, and Day 56.
  The purpose of this arm is to provide a baseline for evaluating the safety and immunogenicity outcomes of QTP101 by comparing the incidence of adverse events (AEs) and immune responses against those observed in the experimental groups. This group includes individuals without prior TB infection, as indicated by their QFT-negative status, and is essential for assessing the specific effects of the investigational vaccine.
  Interventions: Biological: Placebo
- BCG-vaccinated, HIV-negative, QFT-negative and older adults (65-74) with a low dose of QTP101 (Experimental): This study arm evaluates the safety and immunogenicity of a low dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-negative older adults aged 65-74. Participants receive 2 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56.
  This arm focuses on individuals without prior TB infection, as indicated by their QFT-negative status. The primary objective is to assess the safety profile, including adverse events (AEs), and to explore the vaccine's immunogenicity through antibody titers and cytokine responses. The findings will provide key data on the vaccine's effects in older, previously uninfected populations.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-negative and older adults (65-74) with a high dose of QTP101 (Experimental): This study arm investigates the safety and immunogenicity of a high dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-negative older adults aged 65-74. Participants receive 10 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56.
  The arm focuses on individuals without prior TB infection, as indicated by their QFT-negative status. The primary aim is to evaluate the safety profile, including adverse events (AEs), and to assess the immunogenicity of the high-dose vaccine through antibody titers and cytokine production. The findings will help determine the vaccine's suitability and dose optimization for older populations.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-negative and older adults (65-74) with the placebo (Placebo Comparator): This study arm serves as a placebo comparator for BCG-vaccinated, HIV-negative, QFT-negative older adults aged 65-74. Participants receive intramuscular injections of sterile normal saline (placebo) on Day 0, Day 28, and Day 56.
  The purpose of this arm is to establish a baseline for safety and immunogenicity assessments by comparing the incidence of adverse events (AEs) and immune responses against those observed in the experimental groups. This group includes individuals without prior TB infection, as indicated by their QFT-negative status, and plays a crucial role in evaluating the specific effects of the investigational vaccine.
  Interventions: Biological: Placebo
- BCG-vaccinated, HIV-negative, QFT-positive and middle-aged adults (55-64) with a low dose of QTP101 (Experimental): This study arm evaluates the safety and immunogenicity of a low dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-positive middle-aged adults aged 55-64. Participants receive 2 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56.
  This arm targets individuals with prior latent or resolved TB infection, as indicated by their QFT-positive status. The primary objective is to assess the safety profile, focusing on adverse events (AEs), and to explore the vaccine's immunogenicity through antibody titers and cytokine responses. The results will provide valuable data on the vaccine's performance in previously exposed middle-aged adults.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-positive and middle-aged adults (55-64) with a high dose of QTP101 (Experimental): This study arm investigates the safety and immunogenicity of a high dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-positive middle-aged adults aged 55-64. Participants receive 10 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56.
  This arm focuses on individuals with prior latent or resolved TB infection, as indicated by their QFT-positive status. The primary goal is to assess the safety profile, including adverse events (AEs), and to evaluate the immunogenicity of the high-dose vaccine by measuring antibody titers and cytokine responses. The findings will inform dose optimization and vaccine effectiveness in previously exposed middle-aged adults.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-positive and middle-aged adults (55-64) with the placebo (Placebo Comparator): This study arm serves as a placebo comparator for BCG-vaccinated, HIV-negative, QFT-positive middle-aged adults aged 55-64. Participants receive intramuscular injections of sterile normal saline (placebo) on Day 0, Day 28, and Day 56.
  The purpose of this arm is to establish a baseline for evaluating the safety and immunogenicity outcomes of QTP101 in individuals with prior latent or resolved TB infection, as indicated by their QFT-positive status. This comparison will help identify the specific effects of the investigational vaccine by contrasting it with the placebo group in terms of adverse events (AEs) and immune responses.
  Interventions: Biological: Placebo
- BCG-vaccinated, HIV-negative, QFT-positive and older adults (65-74) with a low dose of QTP101 (Experimental): This study arm evaluates the safety and immunogenicity of a low dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-positive older adults aged 65-74. Participants receive 2 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56.
  This arm targets individuals with prior latent or resolved TB infection, as indicated by their QFT-positive status. The primary objective is to assess the safety profile, focusing on adverse events (AEs), and to explore the vaccine's immunogenicity through antibody titers and cytokine responses. The findings will provide critical insights into the vaccine's safety and effectiveness in previously exposed older populations.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-positive and older adults (65-74) with a high dose of QTP101 (Experimental): This study arm investigates the safety and immunogenicity of a high dose of QTP101 in BCG-vaccinated, HIV-negative, QFT-positive older adults aged 65-74. Participants receive 10 μg of ID93 and 5 μg of GLA-SE via intramuscular injection on Day 0, Day 28, and Day 56.
  This arm focuses on individuals with prior latent or resolved TB infection, as indicated by their QFT-positive status. The primary goal is to assess the safety profile, including adverse events (AEs), and to evaluate the vaccine's immunogenicity through antibody titers and cytokine responses. The results will inform dose optimization and effectiveness of the vaccine in older adults with prior TB exposure.
  Interventions: Biological: QTP101
- BCG-vaccinated, HIV-negative, QFT-positive and older adults (65-74) with the placebo (Placebo Comparator): This study arm serves as a placebo comparator for BCG-vaccinated, HIV-negative, QFT-positive older adults aged 65-74. Participants receive intramuscular injections of sterile normal saline (placebo) on Day 0, Day 28, and Day 56.
  The purpose of this arm is to establish a baseline for evaluating the safety and immunogenicity of QTP101 in individuals with prior latent or resolved TB infection, as indicated by their QFT-positive status. Comparing this group to the experimental arms will help identify the specific effects of the investigational vaccine in terms of adverse events (AEs) and immune responses.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: QTP101 — QTP101 consists of ID93 and GLA-SE. ID93 is a recombinant protein antigen comprising four antigens from Mycobacterium tuberculosis (Mtb). The adjuvant GLA-SE is a TLR4 agonist in a stable oil-in-water emulsion.
  Arms: BCG-vaccinated, HIV-negative, QFT-negative and middle-aged adults (55-64) with a high dose of QTP101; BCG-vaccinated, HIV-negative, QFT-negative and middle-aged adults (55-64) with a low dose of QTP101; BCG-vaccinated, HIV-negative, QFT-negative and older adults (65-74) with a high dose of QTP101; BCG-vaccinated, HIV-negative, QFT-negative and older adults (65-74) with a low dose of QTP101; BCG-vaccinated, HIV-negative, QFT-positive and middle-aged adults (55-64) with a high dose of QTP101; BCG-vaccinated, HIV-negative, QFT-positive and middle-aged adults (55-64) with a low dose of QTP101; BCG-vaccinated, HIV-negative, QFT-positive and older adults (65-74) with a high dose of QTP101; BCG-vaccinated, HIV-negative, QFT-positive and older adults (65-74) with a low dose of QTP101
Biological: Placebo — Sterile 0.9% normal saline
  Arms: BCG-vaccinated, HIV-negative, QFT-negative and middle-aged adults (55-64) with the placebo; BCG-vaccinated, HIV-negative, QFT-negative and older adults (65-74) with the placebo; BCG-vaccinated, HIV-negative, QFT-positive and middle-aged adults (55-64) with the placebo; BCG-vaccinated, HIV-negative, QFT-positive and older adults (65-74) with the placebo

SUMMARY:
The purpose of this study is to evaluate the safety and explore the immunogenicity of ID93+GLA-SE compared to placebo following three intramuscular (IM) injections on Days 0, 28 and 56 in the Bacillus Calmette-Guérin (BCG)-vaccinated older adults aged 55 to 74 with negative or positive result on the QuantiFERON-TB (QFT) test. Eligible participants will be randomly assigned based on age group and the QFT test results to receive either QTP101 (Dose 1 and Dose 2) or placebo.

Safety and immunogenicity will be monitored from the first dose until 12 months after the final dose of the investigational product. Blood samples for immunogenicity analysis will be collected at five-time points: before the first dose (Day 0), 4 weeks after the first dose (Day 28), 4 weeks after the second dose (Day 56), 4 weeks after the third dose (Day 84), and 48 weeks after the third dose (Day 392). Once the safety and immunogenicity follow-up is completed 48 weeks after the third dose (Day 392) for the last enrolled participant, a final report will be compiled based on the collected data.

DETAILED DESCRIPTION:
This Phase 1 randomized, double-blind, placebo-controlled clinical trial aims to evaluate the safety and explore the immunogenicity of the investigational tuberculosis (TB) vaccine candidate QTP101 (ID93+GLA-SE) in healthy and medically stable older adults aged 55-74 years. The study targets two specific age groups-55-64 years (middle-aged) and 65-74 years (elderly)-to address the unmet need for effective TB prevention in populations with high disease prevalence and risk, particularly in countries with an aging population.

The trial involves three treatment arms:

Low-dose vaccine group: 2 μg ID93 + 5 μg GLA-SE High-dose vaccine group: 10 μg ID93 + 5 μg GLA-SE Placebo group: Normal saline (0.9%)

Participants will receive three intramuscular (IM) injections of their assigned treatment at baseline (Day 0), Day 28, and Day 56. They will be monitored for safety and immunogenicity over 12 months, with regular follow-up visits scheduled at 1, 6, and 12 months post-final injection.

Key Study Elements:

Eligibility Criteria: Participants must be BCG-vaccinated, HIV-negative, and have QuantiFERON-TB Gold (QFT) test results positive or negative. Chronic conditions are permissible if well-controlled. Women of childbearing potential and men must use approved contraception methods during the study.

Safety Monitoring: Adverse events (AEs) will be closely monitored, categorized as immediate AEs (within 30 minutes of vaccination), solicited local/systemic AEs (within 7 days), unsolicited AEs (up to 28 days), and serious AEs (SAEs) monitored until 12 months post-final dose.

Immunogenicity Assessments: Blood samples will be collected pre-vaccination and at multiple intervals (Day 28, 56, 84, and 392) to measure ID93-specific antibody titers (ELISA) and Th1 cytokine responses (ICS).

Sentinel Design for Older Adults: To ensure participant safety, a sentinel group design is employed for cohorts aged 65-74. Initial vaccination will proceed sequentially within smaller sentinel subgroups, with further cohort enrollment contingent on DSMB approval after reviewing safety data.

Study Objective:

This trial aims to establish the safety profile and preliminary immunogenicity of QTP101 as a step toward addressing the persistent global burden of TB, particularly in vulnerable older populations. The results will inform subsequent clinical development phases to optimize the vaccine's dosing and application.

The study's results will provide critical insights into TB vaccine strategies for aging populations, ensuring a foundation for broader preventative interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who can comply with all scheduled assessment visits during the clinical trial period and who can be continuously monitored by the investigator through the provided contact information
2. Males or females aged 55 to 74 years at the time of consent
3. Participants and/or legally authorized representatives who are capable of providing written informed consent (signed in person in the presence of a witness)
4. Participants with either positive or negative QFT test results at the time of screening; QFT testing can be omitted in the following case: If participants have a documented history of a positive QFT test result, evidenced by submitted records or recorded in the EMR
5. Participants with negative HIV test results at the time of screening
6. Participants with a record of BCG vaccination or BCG scar directly
7. Participants who fall within the following range in physical measurements at the time of screening: 19 ≤ Body Mass Index (BMI) ≤ 33 (kg/m^2) BMI and weight results are rounded to the nearest whole number.
8. Healthy participants or those with well-managed chronic diseases through medical history and clinical examination
9. Female participants must provide evidence at the screening visit (Visit 1) that they meet one of the following criteria to be considered non-fertile:

   * Non-fertile: Defined as post-menopausal or other infertility conditions. Post-menopausal women: No menstrual periods for at least 12 months after stopping all external hormone treatments and over 55 years old. Documented irreversible surgical infertility such as hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. However, tubal ligation is not permitted.
   * Fertile: Women of childbearing potential who have not undergone sterilization must agree to use appropriate contraception during the investigational product administration period and for 6 months after the end of the investigational product administration. They must undergo a serum pregnancy test (β-hCG test) at the screening visit (Visit 1) and urine pregnancy tests (Urine-hCG test) at subsequent visits, with negative HCG results required.
10. Male participants can be enrolled under the following conditions: Men who have not undergone vasectomy must agree to use barrier contraception (e.g., condoms) and agree that both they and their partner will use appropriate contraception during the investigational product administration period and for 6 months after the end of the investigational product administration.
11. Participants who understand the clinical trial procedures, voluntarily decide to participate and sign the informed consent form
12. Participants recommended for tuberculosis prevention treatment who have been adequately informed about and understand latent tuberculosis chemoprophylaxis, and voluntarily agree to participate in the clinical trial while expressing non-consent to the chemoprophylaxis

Exclusion Criteria:

Participants who meet any of the following criteria must be excluded from enrollment.

1. Participants who are suspected of having tuberculosis, have a history of tuberculosis, are currently undergoing treatment for tuberculosis, are being treated for latent tuberculosis infection, or have a history of medication treatment for latent tuberculosis infection at the time of the Screening (Visit 1) or the first administration (Visit 2)
2. Participants who have received other investigational products or used unapproved drugs within 6 months prior to participating in the clinical trial or who plan to use them during the trial period
3. Participants who have previously received an investigational tuberculosis vaccine
4. Participants who test positive for HIV at the screening visit
5. Participants who test positive for HCV or who test positive for HBsAg and negative for HBsAb in HBV tests at the screening visit
6. Participants who are exposed to or will be exposed to investigational or non-investigational products during the clinical trial period or who participate in another clinical trial simultaneously
7. Participants who have received immunoglobulins and/or any blood products within 90 days before the first administration of the investigational product or plan to receive them during the clinical trial period
8. Pregnant or breastfeeding female
9. Participants with the following medical or psychiatric conditions that make it impossible to conduct the clinical trial as judged by the principal investigator:

   * Participants with acute fever (an arbitrary body temperature of 38°C or higher at the time of randomization or within 24 hours before randomization), acute respiratory disease, or active infection.
   * Participants with malignancies or a history of malignancies within the past 5 years.
   * Participants with respiratory diseases: who have received treatment for acute exacerbation or moderate exacerbation of a respiratory condition within 2 years prior to the first administration of the investigational product. (Participants with a history of high-risk pulmonary diseases, such as silicosis, may be excluded at the investigator's discretion, regardless of the treatment period or even if the history is beyond the past 2 years. However, participants with controlled asthma or COPD stage 0 (at-risk) may participate with judgment of the principal investigator.)
   * Participants with serious cardiovascular diseases: congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension, etc.
   * Participants with neurological diseases: epilepsy, seizures within 3 years before the first administration of the investigational products, migraines, strokes, encephalopathy, Guillain-Barre syndrome, etc.
   * Participants with a history of COVID-19 infection within 90 days before the screening visit (confirmed positive by NAAT or rapid antigen test) or who have not recovered from COVID-19-related symptoms after being diagnosed with COVID-19 more than 90 days before the screening visit.
   * Participants with autoimmune hypothyroidism, autoimmune diseases, immunodeficiency diseases.
   * Participants with other clinically significant medical histories related to the hepatobiliary system, kidneys, endocrine system, urinary system, musculoskeletal system, etc., as judged by the principal investigator.
   * Participants with a history of hereditary or idiopathic angioedema.
   * Participants with a history of organ or bone marrow transplantation.
   * Participants with a history of platelet-related or bleeding disorders, a history of significant bleeding or bruising following intramuscular injection or venipuncture, or who are receiving anticoagulants.
10. Participants who have received radiation therapy within 12 months before the first administration of the investigational product. However, those who have received radiation therapy to the lungs are excluded regardless of the time frame.
11. Participants who have surgery planned during the clinical trial period
12. Participants with a history of severe allergic reactions or anaphylaxis to vaccines or other allergens
13. Participants with clinically significant abnormal findings in laboratory tests, ECG, or chest X-ray at the screening visit as judged by the principal investigator to be unsuitable for participation. Participants with fibrotic nodular lesions on chest X-ray (indicative of spontaneously healed tuberculosis lesions without a history of tuberculosis treatment)
14. Participants who have chronically received immunosuppressants or other immunomodulatory drugs within 6 months before the first administration of the investigational product

    * High-dose corticosteroids (continuous use of doses exceeding 15 mg/day of prednisolone for more than 14 days)
    * However, topical steroids, nasal sprays, inhalers, and eye drops are allowed regardless of the dose
15. Participants who are deemed unsuitable for this clinical trial by the principal investigator for any other reasons
16. Participants with cognitive impairment.
17. Household contacts and close contacts who have been in an indoor environment with an active tuberculosis patient

    * Household Contact: Family members and cohabitants who have been living in the same space or regularly interacting for at least 3 months.
    * Close Contact: Individuals other than household contacts who have had direct contact in an enclosed indoor environment (e.g., classroom, office) for an extended period, defined as continuous or daily contact for at least 8 hours per day, or cumulative contact of 40 hours or more.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint - Immediate Adverse Events | Within 30 minutes after each administration
  Immediate adverse events within 30 minutes after administration
Safety Endpoint - Solicited local and systemic Adverse Events | Occurred up to 7 days after each administration
  Solicited local/systemic AEs occurred up to 7 days after administration
Safety Endpoint - Unsolicited local and systemic Adverse Events | Occurred up to 28 days after each administration
  Unsolicited local/systemic AEs occurred up to 28 days after administration
Safety Endpoint - Serious Adverse Events and Adverse Event of of Special Interest | Occurred from the first administration up to 48 weeks after the last administration
  Serious AE (SAEs) and AE of special interest (AESI) occurred from the first administration up to 48 weeks after the last administration
Safety Endpoint - Laboratory assessment (Hematological Test) | From screening to the end of visit at 48 weeks after the last administration
  Hematological test for each participant
Safety Endpoint - Laboratory assessment (Hematochemical test) | From screening to the end of visit at 48 weeks after the last administration
  Hematochemical test for each participant
Safety Endpoint - Laboratory assessment (Urine test) | From screening to the end of visit at 48 weeks after the last administration
  Urine test for each participant
Safety Endpoint - Vital Signs (Body temperature) | From screening to the end of visit at 48 weeks after the last administration
  Body weight will be measured at each scheduled visit after the administration of the investigational product for each participant.
Safety Endpoint - Vital Signs (Pulse) | From screening to the end of visit at 48 weeks after the last administration
  Pulse rate will be measured for each participant.
Safety Endpoint - Vital Signs (Respiratory rate) | From screening to the end of visit at 48 weeks after the last administration
  Respiratory rate will be measured for each participant.
Safety Endpoint - Vital Signs (Blood pressure) | From screening to the end of visit at 48 weeks after the last administration
  Systolic and diastolic blood pressure will be measured for each participant.
Immunogenicity Endpoint - Humoral immunity (GMT) | Before 1st administration, 4 weeks after 1st administration, 4 weeks after 2nd administration, 4 and 48 weeks after 3rd administration
  Geometric mean titer (GMT) of antigen-specific IgG measured with ELISA
Immunogenicity Endpoint - Humoral immunity (GMFR) | Before 1st administration, 4 weeks after 1st administration, 4 weeks after 2nd administration, 4 and 48 weeks after 3rd administration
  Geometric mean fold rise (GMFR) of antigen-specific IgG measured with ELISA
Immunogenicity Endpoint - Humoral immunity (SRR) | Before 1st administration, 4 weeks after 1st administration, 4 weeks after 2nd administration, 4 and 48 weeks after 3rd administration
  Seroresponse rate (SRR), defined as a 4-fold rise in antibody titer of antigen-specific IgG measured with ELISA from Baseline
Immunogenicity Endpoint - Cellular immunity (ICS) | Before 1st administration, 4 weeks after 1st administration, 4 weeks after 2nd administration, 4 and 48 weeks after 3rd administration
  The ratio and amount of antigen-specific Th1 cytokine-secreting cells measured with intracellular cytokine staining (ICS)
Immunogenicity Endpoint - Cellular immunity (RR) | Before 1st administration, 4 weeks after 1st administration, 4 weeks after 2nd administration, 4 and 48 weeks after 3rd administration
  Cell response rate (RR), defined as a 4-fold rise in the amount of antigen-specific Th1 cytokine-secreting cells from the baseline.
Safety Endpoint - Physical examinations (General Appearance) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Overall health and appearance, including posture and obvious abnormalities.
Safety Endpoint - Physical examinations (Skin) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Inspection for rashes, lesions, discoloration, or other visible skin issues
Safety Endpoint - Physical examinations (Head/Neck) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Examination of the skull, scalp, lymph nodes, and thyroid gland
Safety Endpoint - Physical examinations (Chest/Lungs) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Assessment of respiratory sounds, chest wall movement, and breathing patterns using inspection and auscultation
Safety Endpoint - Physical examinations (Heart) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Evaluation of heart sounds, rhythm, and potential murmurs through auscultation and palpation
Safety Endpoint - Physical examinations (Abdomen) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Palpation and auscultation for organ enlargement, tenderness, or abnormal bowel sounds
Safety Endpoint - Physical examinations (Genitourinary System) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Examination of genital and urinary organs, focusing on abnormalities or patient-reported symptoms (if applicable)
Safety Endpoint - Physical examinations (Limbs) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Inspection and assessment for swelling, deformities, or movement limitations
Safety Endpoint - Physical examinations (Musculoskeletal System) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Examination of joints, muscles, and bones for pain, swelling, or restricted mobility
Safety Endpoint - Physical examinations (Nervous System) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Assessment of reflexes, motor and sensory functions, and coordination
Safety Endpoint - Physical examinations (Other) | At screening, the second and third administrations, 4, 24 and 48 weeks after the last administration.
  Any additional assessments based on the participant's symptoms or clinical findings

CONTACTS AND LOCATIONS:
Overall Officials: Jinhee Lee, DVM, PhD, Study Director — Quratis Inc.; Jae Chol Choi, MD, PhD, Principal Investigator — Chung-Ang University Gwangmyeong Hospital; Youngmok Park, MD, PhD, Principal Investigator — Severance Hospital; Kwang Joo Park, MD, PhD, Principal Investigator — Ajou University School of Medicine; Jinsoo Min, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (4):
- South Korea (4):
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong, Gyeonggi-do
  - Yonsei University Severance Hospital, Seoul
  - The Catholic University of Korea Seoul ST.MARY'S Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared for research purposes through publication in peer-reviewed journals. The data will be presented in aggregate form or as part of supplementary materials accompanying the manuscript, ensuring participant confidentiality through anonymization.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available following the publication of the study results in peer-reviewed journals. This is expected within [specify timeframe, e.g., 6 months to 1 year] after the completion of the study.
Access Criteria: Access to the data will be limited to the information published in peer-reviewed journals. Additional data requests beyond the published information may be considered upon reasonable request and subject to institutional and ethical approvals.